CLINICAL TRIAL: NCT01048944
Title: NRT & Bupropion Mechanisms of Effectiveness in Smokers: Phase IV Trial
Brief Title: Nicotine Replacement Therapy (NRT) and Bupropion Mechanisms of Effectiveness in Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern Illinois University Carbondale (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Gilbert, Professor of Psychology, Southern Illinois University Carbondale
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: NIH/NIDA-2R01DA012289; 2R01DA012289 (NIH)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Nicotine Dependence
Keywords: Electroencephalography; nicotine; bupropion; attention; drug withdrawal symptoms
MeSH Terms: conditions — Tobacco Use Disorder; Substance Withdrawal Syndrome | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bupropion SR (Active Comparator): 150 mg bid bupropion SR
  Interventions: Drug: Bupropion SR
- Nicotine Patch (Active Comparator): 21mg, 14mg, 7mg
  Interventions: Drug: Nicotine Patch
- Placebo Patch and Placebo Pill (Placebo Comparator): Individuals were placed on both a placebo patch that were the same size as active patches given to the Nicotine Patch group and were also given placebo pills were the same size and identically packaged as the active pills (bupropion) given to the Bupropion SR group.
  Interventions: Drug: Placebo Patch and Placebo Pill
- Delayed-quit control (No Intervention): Smoke for 67 days while others have quit, then quit.

INTERVENTIONS:
Drug: Bupropion SR — 150 encapsulated pill,3 days 1x/day then 56/day for 2x/day, then 3 day 1x/day ramp-down.
  Other Names: ZybanSR
  Arms: Bupropion SR
Drug: Nicotine Patch — Nicotine patch beginning 1st day cessation: 21 mg/24 days, 14 mg/14 days, 7 mg/7 days
  Other Names: NicodermCQ
  Arms: Nicotine Patch
Drug: Placebo Patch and Placebo Pill — 150 encapsulated placebo pill,3 days 1x/day then 56/day for 2x/day, then 3 day 1x/day ramp-down. Placebo patch beginning 1st day cessation: 21 mg/24 days, 14 mg/14 days, 7 mg/7 days. The placebo patches were given beginning 1st day cessation: 21 mg size (but actually placebo)/24 days, 14 mg size (actually placebo)/ 14 mg size (actually placebo) 14 days/, 7 mg size (actually placebo)/7 days
  Other Names: Placebo
  Arms: Placebo Patch and Placebo Pill

SUMMARY:
The purpose of this study is to better characterize differences in mood, attention, brain activation patterns underlying the beneficial effects of pharmacological treatments previously demonstrated to be help individuals successfully quit tobacco smoking. Smokers will be randomly assigned to one of three treatments: 1) bupropion sustained release (SR), 2) nicotine patch, or 3) placebo patches plus pills across a 45-day period with a 3-week intensive post-treatment follow-up. In addition, 20 percent of the subjects will be randomized to a delayed-quit control group.

DETAILED DESCRIPTION:
The first aim of this revised proposal is to accurately assess the duration and trajectories of smoking abstinence symptoms and associated biobehavioral indices across 66 days of quitting smoking in 3 different treatment groups: 1) bupropion SR (BUP), 2) transdermal nicotine patch (TNP), and 3) placebo patch plus placebo pill. Study sensitivity and accuracy will be maximized by using procedures designed to maximize abstinence and minimize study dropout. The second aim is to characterize brain and psychological mechanisms by which BUP and TNP promote abstinence. While the efficacies of BUP and TNP in promoting smoking abstinence have been repeatedly demonstrated, little is known about the mechanisms mediating this efficacy. The final primary goal of this competitive continuation proposal is to characterize individual differences in psychological and brain mechanisms mediating the beneficial effects of BUP and TNP on smoking abstinence and withdrawal symptoms. A secondary goal is to assess the ability of a battery of innovative brain and biobehavioral measures of attention and affect to predict relapse.

To achieve these goals, the effects of quitting smoking with or without the help of TNP and BUP will be assessed intensively across 66 days of abstinence. Dependent measures will be mood, vigilance, attentional bias to smoking and emotional stimuli, and related physiological measures (resting EEG activation and activation asymmetry indices of affective states and traits, and event-related potential activity elicited by emotional and smoking stimuli). Smokers will be randomly assigned to one of three immediate-quit groups (N = 60 per group): (1) bupropion + placebo patch, (2) placebo pill + nicotine patch, and (3) placebo patch + placebo pill; or to a fourth (control) group (N = 40) that will quit after the final experimental session (after the other subjects have completed their 66-day* abstinence period). Subjects in the 3 treatment groups and the control group will have the same set of biobehavioral measures assessed during the experimental sessions at the same points in time. It is hypothesized that BUP and TNP will have both common and unique mechanisms by which they reduce withdrawal symptoms and that gender and personality traits will moderate the effects of these treatments. (Note.* To avoid final-session mood and arousal effects subjects will actually quit for 67 days, but biobehavioral measures will be collected on the 66th day of abstinence.)

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Diagnostic and Statistical Manual of the American Psychiatric Association (DSM-IV) diagnosis of nicotine dependence with psychological dependence
* Smokes at least 10 cigarettes per day for the three months prior to enrollment
* Currently seeking treatment for nicotine dependence
* Medically healthy on the basis of physical examination and medical history, vital signs,
* Females must use an effective method of contraception for the duration of the study

Exclusion Criteria:

* DSM-IV diagnosis of abuse or dependence on alcohol or drugs other than nicotine
* Current Axis I diagnosis or current treatment with psychotropic medications within the three months prior to enrollment
* History of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders
* Currently seeking treatment for nicotine disorders
* History of seizures or head trauma with loss of consciousness, brain contusion, or fracture
* History of significant recent violent behavior
* Blood pressure greater than 150/90
* History of eating disorders
* History of allergic reaction to any of the study medications
* Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2005-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Gilbert, PhD, Principal Investigator — Southern Illinois University Carbondale
Locations (1):
- Southern Illinois University, Carbondale, Illinois, United States

REFERENCES:
- [Derived] Gilbert DG, Rabinovich NE, Gilbert-Matuskowitz EA, Klein KP, Pergadia ML. Smoking abstinence symptoms across 67 days compared with randomized controls-Moderation by nicotine replacement therapy, bupropion, and negative-affect traits. Exp Clin Psychopharmacol. 2019 Dec;27(6):536-551. doi: 10.1037/pha0000278. Epub 2019 Mar 28. PMID 30920255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: 9/01/06 to 9/01/11. Recruitment was throughout Carbondale and surrounding communities and occurred with newspaper ads, flyers, radio and television presentations. Recruitment was more challenging than expected because of the large time commitment and high prevalence of psychoactive medication and drug use (exclusionary criteria).
Pre-assignment Details: After consent subjects and the completion of their first experimental session subjects were randomly assigned to one of 4 treatment arms: 197 signed the consent, 126 completed the first experimental session and were subsequently randomly assigned to a treatment condition.
Groups:
- Bupropion Sustained Release (SR): 150 mg bid bupropion SR
  Bupropion SR: 150 encapsulated pill,3 days 1x/day then 56/day for 2x/day, then 3 day 1x/day ramp-down.
- Nicotine Patch: 21mg, 14mg, 7mg
  Nicotine: Nicotine patch beginning 1st day cessation: 21 mg/24 days, 14 mg/14 days, 7 mg/7 days
- Placebo Patch and Placebo Pill: Placebo patch same size as active patches
  Placebo pill and Placebo Patch: 150 encapsulated placebo pill,3 days 1x/day then 56/day for 2x/day, then 3 day 1x/day ramp-down. Placebo patch beginning 1st day cessation: 21 mg/24 days, 14 mg/14 days, 7 mg/7 days.
Period: Overall Study
Arm/Group | Bupropion Sustained Release (SR) | Nicotine Patch | Placebo Patch and Placebo Pill | Delayed-quit Control
Started | 32 | 38 | 35 | 21
Completed | 24 | 28 | 25 | 19
Not Completed | 8 | 10 | 10 | 2
Not completed — Protocol Violation | 8 | 10 | 10 | 2

BASELINE CHARACTERISTICS:
Population: Personality trait questionnaires, history of psychiatric disorders, SES, age, smoking and drug use history.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion SR | Nicotine Patch | Placebo Patch and Placebo Pill | Delayed-quit Control | Total
Number analyzed (Participants) | 32 | 38 | 35 | 21 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.85 (11.76) | 30.84 (11.00) | 31.49 (10.44) | 26.8 (10.42) | 30.64 (10.97)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 1 | 2 | 7
  Between 18 and 65 years | 30 | 36 | 34 | 19 | 119
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 18 | 8 | 58
  Male | 18 | 20 | 17 | 13 | 68
Region of Enrollment [Number; unit: participants]
  United States | 32 | 38 | 35 | 21 | 126

OUTCOME MEASURES:

1. Primary Outcome: Changes in Log Brain-wave (EEG) Activity (Power [Microvolts Squared]) From Pre-quit Baseline to 66 Days Post-quit, Assessed at 3, 24, 45, and 66 Days Post-quit.
Description: Brain-wave activity (EEG) was assessed using electrodes on the subject's scalp, the outputs of which were and quantified by a commercial brain wave machine. EEG was collected at frontal (e.g., Fz) and parietal (e.g., Pz) electrodes while subjects relaxed. EEG was analyzed using computer programs that measured slow-frequency EEG waves known as delta (1.5-4.5 cycles/second [cps]), theta-1 (4.5-6.0 cps), theta-2 (6.0-7.7 cps), and alpha-1 (7.8-10.0 cps), and higher frequency waves. Generally, delta, alpha-1 and theta waves reflect deactivation of the brain activity, while higher frequency waves reflect greater brain activation. Brain activity was quantified as the natural log of EEG power [microvolts squared] as determined by the fast Fourier mathematical algorithm. Days post quit were components of Time. The primary focus was on changes in the individual subject's log theta-1, theta-2, and alpha-1 power at post-quit points in time minus the log values at the pre-quite baseline.
Time Frame: Mean EEG power [microvolts squared] from at baseline, 3, 24, 45, and 66 days post-quit
Population: For the currently reported analyses, only individuals complying with the study requirements, including biochemically verified smoking abstinence, were assessed. Future analyses will include individuals who complied to certain critical endpoints.
Measure: Mean (Standard Error); unit: Change in log EEG [microvolts squared]
Arm/Group | Nicotine Patch | Bupropion SR | Placebo Patch and Placebo Pill | Delayed-quit Control
Number analyzed (Participants) | 28 | 24 | 25 | 19
Change in log EEG [microvolts squared]
  Day-3 Change in log Theta-1 EEG Power Fz | .055 (.061) | .224 (.066) | .234 (.066) | -.094 (.071)
  Day-24 Change in log Theta-1 EEG Power Fz | .194 (.068) | .198 (.074) | .258 (.074) | -.060 (.080)
  Day-45 Change in log Theta-1 Power Fz | .232 (.055) | .249 (.060) | .161 (.060) | -.032 (.065)
  Day-66 Change in log Theta-1 EEG Power Fz | .431 (.075) | .407 (.081) | .184 (.081) | -.026 (.087)
  Day-3 Change in log Theta-2 Power Fz | .062 (.077) | .088 (.083) | .249 (.083) | -.070 (.090)
  Day-24 Change in log Theta-2 Power Fz | .251 (.087) | .150 (.094) | .278 (.094) | -.042 (.101)
  Day-45 Change in log Theta-2 Power Fz | .319 (.074) | .248 (.081) | .278 (.094) | .054 (.087)
  Day-66 Change in log Theta-2 Power Fz | .504 (.092) | .502 (.100) | .205 (.100) | .001 (.107)
  Day-3 Change in log Alpha-1 Power Pz | -.023 (.103) | .155 (.112) | .184 (.112) | -.004 (.121)
  Day-24 Change in log Alpha-1 Power Pz | .139 (.099) | .301 (.107) | .276 (.107) | -.001 (.115)
  Day 45 Change in log Alpha-1 Power Pz | .292 (.099) | .261 (.107) | .259 (.107) | .021 (.115)
  Day 66 Change in log Alpha-1 Power Pz | .339 (.099) | .459 (.107) | .292 (.107) | .017 (.116)
Statistical Analysis 1: Comparison: Nicotine Patch vs Bupropion SR vs Placebo Patch and Placebo Pill vs Delayed-quit Control; Mixed-model repeated measures multivariate analyses of variance assessed Treatment x Day of abstinence (days 3, 24, 45, and 66) based on changes from pre-quit baseline to values of the four post-quit time points (days 3, 24, 45, and 66); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — P values are adjusted for multiple comparisons except for specific a priori directional predictions

2. Primary Outcome: Changes in Log of Smoking Withdrawal Scores (Mood, and Depressive Symptoms) From Baseline Across 66 Days of Abstinence
Description: Changes in log from baseline in the widely used Shiffman-Jarvik Withdrawal "craving" and "psychological symptom" scores through 66 days of abstinence. Post-quit changes were assessed at days 3, 24, 45, and 66 of abstinence. The maximal range of value raw for craving is from "5" = (no craving) to "47" (maximally strong craving), while that for psychological symptoms is from "5" (no symptoms) to "60" (maximally intense symptoms of across multiple symptoms). Because the subtraction of logs is equivalent to the ratio of the two scores, a difference in logs (base 10) with a value of "1" is equal to an increase by a factor of 10, while a value of "0" is no change, and values of less than "0" are decreases below baseline values.
Time Frame: Changes in log withdrawal symptoms from baseline through 66 days of abstinence
Population: Analysis population included only those individuals who complied fully with study requirements through 67 days of abstinence.
Measure: Mean (Standard Error); unit: log (base 10) units on a scale
Arm/Group | Nicotine Patch | Bupropion SR | Placebo Patch and Placebo Pill | Delayed-quit Control
Number analyzed (Participants) | 28 | 24 | 25 | 19
log (base 10) units on a scale
  Day-3 Change in log Shiffman Craving | -.006 (.038) | .045 (.042) | .094 (.040) | -.045 (.046)
  Day-24 Change in log Shiffman Craving | -.187 (.054) | -.199 (.060) | -.045 (.057) | -.059 (.066)
  Day-45 Change in log Shiffman Craving | -.273 (.047) | -.201 (.052) | -.132 (.050) | -.043 (.057)
  Day-66 Change in log Shiffman Craving | -.236 (.054) | -.230 (.059) | -.205 (.057) | -.075 (.065)
  Day-3 Change in log Shiffman Psych Withdrawal | .089 (.032) | .210 (.035) | .172 (.034) | .016 (.039)
  Day-24 Change in log Shiffman Psych W | .065 (.031) | .102 (.034) | .076 (.033) | -.025 (.038)
  Day-45 Change in log Shiffman Psych Withdrawal | .008 (.031) | .063 (.034) | .039 (.033) | -.017 (.038)
  Day-66 Change in log Shiffman Psych Withdrawal | .068 (.037) | .032 (.041) | .029 (.039) | -.012 (.045)

ADVERSE EVENTS:
Time Frame: From the day of consent through one year after the 67-day post-quit treatment phase.
Description: Questionnaires at approximately weekly intervals through one year after the 67-day post-quit treatment phase. Then every 3 months until a year after the study.
Groups:
- Bupropion SR: 150 mg bid bupropion SR
  Bupropion SR: 150 encapsulated pill, 3 days 1x/day then 56 days at 2x/day, then 3 day at 1x/day ramp-down.
- Placebo Patch and Placebo Pill: Placebo patch same size as active patches
  Placebo pill and Placebo Patch: 150 encapsulated placebo pill,3 days 1x/day then 56 days at 2x/day, then 3 days at 1x/day ramp-down. Placebo patch beginning 1st day cessation: 21 mg/24 days, 14 mg/14 days, 7 mg/7 days.
Arm/Group | Bupropion SR | Nicotine Patch | Placebo Patch and Placebo Pill | Delayed-quit Control
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/38 | 0/35 | 0/21
Other Adverse Events (participants affected / at risk) | 21/32 | 22/38 | 19/35 | 6/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion SR (N=32) | Nicotine Patch (N=38) | Placebo Patch and Placebo Pill (N=35) | Delayed-quit Control (N=21)
Dry Mouth (Gastrointestinal disorders) | 13 (53) | 13 (34) | 9 (27) | 2 (2) — Self-reported "dry mouth" on standard questionnaire
Sleep disturbance (Psychiatric disorders) | 13 (42) | 15 (63) | 17 (54) | 2 (6) — Self-reported "sleep disturbance" on standard questionnaire.
Headaches (Nervous system disorders) | 3 (7) | 3 (3) | 3 (4) | 3 (5) — Self-reported "headaches"
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (12) | 2 (3) | 1 (1)
Dizzyness (Nervous system disorders) | 3 (5) | 1 (6) | 5 (7) | 0 (0) — Self-reported "dizziness"

LIMITATIONS AND CAVEATS:
The modest sample size limited the ability to detect more subtle treatment effects. The exclusionary criteria limits generalization to excluded groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No